CLINICAL TRIAL: NCT05890404
Title: Implementing Sustainable Evidence-based Mental Healthcare in Low-resource Community Settings Nationwide to Advance Mental Health Equity for Sexual and Gender Minority Individuals
Brief Title: SGM Evidenced-Based Mental Healthcare Implementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Northwestern University (Other); Arizona State University (Other); Miami University (Other); University of Miami (Other); CenterLink (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000035211; 1R01MH133543-01 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: CBT; LGBTQ

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Materials Only (Experimental): The Materials Only arm will have access to a digital suite of online training materials for LGBTQ-Affirmative CBT prepared by the research team.
  Interventions: Behavioral: LGBTQ-Affirmative CBT Training: Materials Only
- Direct Training (Experimental): In addition to receiving access to the online training materials, the Direct Training arm will receive 12 weekly 1-hour live webinars on delivering LGBTQ-affirmative CBT led by our four expert trainers.
  Interventions: Behavioral: LGBTQ-Affirmative CBT Training: Direct Training
- Local Supervision (Experimental): In addition to receiving the online training materials and live webinars, the Local Supervision arm will receive guidance from an on-site clinical supervisor, who will be nominated by the center director as someone with substantial CBT experience.
  Interventions: Behavioral: LGBTQ-Affirmative CBT Training: Local Supervision

INTERVENTIONS:
Behavioral: LGBTQ-Affirmative CBT Training: Materials Only — Participants will be provided a digital suite of online self-guided learning materials, including step-by-step treatment materials, client handouts, and "how to" instructions for delivering the treatment.
  Arms: Materials Only
Behavioral: LGBTQ-Affirmative CBT Training: Direct Training — Participants will be provided a digital suite of online self-guided learning materials, including step-by-step treatment materials, client handouts, and "how to" instructions for delivering the treatment. In addition, participants will receive 12 weekly 1-hour live training webinars on delivering LGBTQ-affirmative CBT led by expert trainers.
  Arms: Direct Training
Behavioral: LGBTQ-Affirmative CBT Training: Local Supervision — Participants will be provided a digital suite of online self-guided learning materials, including step-by-step treatment materials, client handouts, and "how to" instructions for delivering the treatment. In addition, participants will receive 12 weekly 1-hour live training webinars on delivering LGBTQ-affirmative CBT led by expert trainers. This arm will also receive one year of ongoing (at least monthly) supervision in LGBTQ-affirmative CBT from an expert supervisor at your center.
  Arms: Local Supervision

SUMMARY:
The purpose of the proposed study is to identify effective strategies for implementing lesbian, gay, bisexual, transgender, and queer (LGBTQ)- affirmative Cognitive-Behavioral Therapy (CBT) at LGBTQ community centers across the United States.

DETAILED DESCRIPTION:
The purpose of the proposed study is to identify effective strategies for implementing lesbian, gay, bisexual, transgender, and queer (LGBTQ)-affirmative CBT (cognitive-behavioral therapy) at LGBTQ community centers across the United States. This study will specifically compare the effectiveness of three implementation strategies: (1) training materials only, (2), training materials and direct training from our expert trainers, and (3) training materials, direct training, and local supervision from a clinical supervisor. The proposed prospective study will utilize a type 3 hybrid implementation-effectiveness trial. This design is used to compare the impact of two or more implementation strategies while also gathering effectiveness data and is recommended when there is already strong evidence for the intervention's effectiveness, strong basis that the implementation strategies are feasible, and strong implementation momentum. Randomization will occur on the center-level, so that MHPs working in the same center will receive one of the three types of training.

Outcomes include mental health providers' changes in demonstrated skills in providing LGBTQ-affirmative CBT from baseline to 4-, 8-, 12-, and 24-months post-baseline. This study will also investigate determinants of successful implementation of LGBTQ-affirmative CBT and examine the impact of the implementation strategies on client mental health.

ELIGIBILITY:
Inclusion Criteria: Providers

Eligible providers will meet the following criteria:

* 18 years of age or older
* working as a psychologist, psychiatrist, social worker, mental health counselor, nurse practitioner, or peer support provider
* affiliated with a US LGBTQ community center
* providing mental health services to at least one sexual or gender minority (SGM) client

Exclusion Criteria: Providers

Providers will be deemed ineligible due to:

- possessing substantive experience with LGBTQ-affirmative CBT (e.g., having read most the LGBTQ-affirmative CBT treatment manual, attended LGBTQ-affirmative CBT training, or been supervised by someone who has previously attended the LGBTQ-affirmative CBT training)

Inclusion Criteria: Clients

Eligible clients will meet the following criteria:

* of age to consent to mental health treatment in the state in which they live
* receiving ongoing mental health services at one of the 15 LGBTQ centers selected for the client evaluation aim of the present study
* self-identifying as LGBTQ

Exclusion Criteria: Clients

There are no exclusion criteria for clients

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Provider Implementation Fidelity | 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Provider implementation fidelity of LGBTQ-Affirmative Therapy will serve as the primary implementation outcome and will be measured using a simulated practice assessment. Providers will watch two brief (three-minute) video clips of an SGM actor roleplaying a presenting concern and briefly describe in writing the clinical approaches they would use to address the concern. Research assistants will code the videos for important themes using a a scale created by expert LGBTQ-affirmative trainers for this study. This 2-item Likert scale ranges from 0 (did not mention [theme]) to 2 (discussed [theme] in-depth), and has a score range of 0-4. A higher score is indicative of a higher fidelity to the the treatment protocol. Administration time is 20 minutes.
Change in Client Depression Symptoms | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client depression symptoms will serve as the primary effectiveness outcome and will be Client depression symptoms will be measured on the client survey using the 9-item version of the Patient Health Questionnaire (PHQ-9). Participants respond to each item on a scale of 0 ("not at all") to 3 ("nearly every day"). Total scores range from 0-27, and are calculated as the sum of the 9 items. A higher score of indicative of higher depression symptomatology. Administration time is 6 minutes.

SECONDARY OUTCOMES:
Change in Reach of LGBTQ-affirmative CBT. | 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Reach of LGBTQ-affirmative CBT will be assessed on the provider survey as the percent of clients who receive LBGTQ-affirmative CBT out of total center clients. Total scores range from 0-100%; a higher percent indicates a stronger reach of LGBTQ-affirmative CBT. Additionally, opened-ended questions in provider interviews will highlight reasons for stronger or weaker reach.
Change in Adoption of LGBTQ-affirmative CBT | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Adoption of LGBTQ-affirmative CBT will be assessed on the provider survey as percent of providers who practice LGBTQ-affirmative CBT out of number trained. The range for this measure is 0-100%. Semi-structured qualitative interviews with providers will highlight why and in what cases providers chose not to implement. We will also use secondary data from CenterLink to describe factors of centers choosing not to receive training.
Change in Familiarity With and Use of LGBTQ-affirmative CBT skills | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Familiarity with and use of LGBTQ-affirmative CBT skills will be assessed on the provider survey using Familiarity and Use Scale. This instrument contains 14 items, to which participants respond to each item on a Likert scale from 1 ("not at all"/"not at all familiar" ) to 5 ("very often"/"extremely familiar").* The total score is calculated by summing the items, and can range from 1-70. A higher score indicates higher familiarity with and use of LGBTQ-affirmative CBT skills. Administration time is 7 minutes.
  *Dependent on the phrasing/context of the item
Change in Modification of LGBTQ-affirmative CBT | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Modification of LGBTQ-affirmative CBT will be assessed on the provider survey using the Modification and Adaptation Checklist. This instrument contains 14 items as well as corresponding codes (0 -12) that denote different types of modifications. As these codes do not have corresponding values, this measure is not scored. Administration time is
Change in Adaptation to Local Contexts and Clients | 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Adaptation to local contexts and clients will be assessed on the provider interview following our published guidance on intentional adaptation to local contexts/clients, as covered in the training.
Change in Maintenance of LGBTQ-affirmative CBT | 4-mo follow-up, 8-mo follow-up, 12-mo follow-up, and 24-mo follow-up
  Maintenance of LGBTQ-affirmative CBT will be assessed on the director survey and provider survey using the Program Sustainability Assessment Tool. This instrument contains 8 subscales and 40 total items, to which participants respond to each item on a Likert scale from 1 ("little or no extent" ) to 7 ("a very great extent"). The total score is calculated by first computing the mean for each subscale, and then computing the means of those scores. The total score can range from 1-7. A higher score indicates stronger maintenance of LGBTQ-affirmative CBT. Administration time is 15 minutes.
  operationalized as ongoing program support, funding stability, center capacity, and fit with strategic planning of LGBTQ-affirmative CBT. Assessed via the director survey and the provider survey and interview.
Change in Client Anxiety | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client anxiety will be assessed on the client survey using Generalized Anxiety Disorder Scale, 7 item Version. Participants respond on a Likert scale from 0 ("not at all") and 3 ("nearly every day"). The total score is calculated by summing the scores for each item, resulting in a range of 0-15. A higher score indicates higher anxiety symptomatology. Administration time is 5 minutes.
Change in Client PTSD Symptoms | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client PTSD symptoms will be measured on the client survey using the PTSD Checklist for Diagnostic and Statistical Manual-5. This instrument contains 20 items, to which participants respond on a Likert scale from 0 ("not at all") to 4 ("extremely") The total score is calculated by summing the scores for each item, resulting in a range of 0-80. A higher score indicates higher PTSD symptomatology. Administration time is 10 minutes.
Change in Client Alcohol Use Behavior | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client alcohol use behavior will be assessed on the client survey using the Alcohol Use Disorders Identification Test - Consumption. This instrument contains 3 items, to which participants respond on a Likert scale from 0 to 4 (the value of each point changes for each question). The total score is calculated by summing the scores for each item, resulting in a range of 0-12. A higher score indicates greater alcohol consumption. Administration time is 2 minutes.
Change in Client Substance Use Behavior | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client substance use* behavior will be assessed on the client survey using the Drug Use Disorders Identification Test - Consumption. This instrument 4 items, to which participants respond on a Likert scale from 0 to 4 (the value of each point changes for each question). The total score is calculated by summing the scores for each item, resulting in a range of 0-16. A higher score indicates greater substance consumption. Administration time is 2 minutes.
  *excluding alcohol
Change in Client internalized stigma | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client internalized stigma will be assessed on the client survey using the 3-item Internalized Stigma subscale of the Lesbian, Gay, Bisexual Identity Scale (LGBIS). Participants respond on a Likert scale from 1 ("disagree strongly" to 6 ("agree strongly"). The total score is calculated by first computing the mean for each subscale, and then computing the means of those scores. The range for possible total scores is 1-18. A higher score indicates greater internalized stigma. Administration time is 2 minutes.
Change in Client Social Isolation | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client social isolation will be assessed on the client survey using the UCLA Loneliness Scale. This instrument contains 3 items, to which participants respond on a Likert scale from 1 ("hardly ever") to 3 ("often"). The total score is calculated by summing the scores for each item, resulting in a range of 1-9. A higher score indicates greater social isolation. Administration time is 2 minutes.
Change in Client Emotion Dysregulation | Baseline, 4-month follow-up, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Client emotion dysregulation will be assessed on the client survey using the Difficulties in Emotion Regulation Scale - Short Form. This instrument contains 6 subscales and 18 total items, to which participants respond on a Likert scale from 1 ("almost never") to 5 ("almost always"). The total score is calculated by summing the scores for each item, resulting in a range of 1-18. A higher score indicates greater difficulties emotional regulation. Administration time is 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale LGBTQ Mental Health Initiative with the Yale School of Public Office, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pachankis JE, Chiaramonte D, Baldwin HT, Prachniak C, Levine DS, Van S, Hobbs RJ, Ankrum H, Wilkins LJ, Harvey TD, Harkness A, Jackson SD, Matsuno E, Soulliard ZA, Last BS, Burger J, Delehant M, Zhou X, Hagaman AK, Li DH, Mustanski B. Implementing LGBTQ-affirmative CBT: study protocol for an effectiveness-implementation trial at 90 LGBTQ community centers. BMC Health Serv Res. 2025 Jul 21;25(1):962. doi: 10.1186/s12913-025-13136-3. PMID 40691571